CLINICAL TRIAL: NCT04054895
Title: LEft VEntricuLar Activation Time Shortening With Physiological Pacing vs Biventricular Resynchronization Therapy: a Randomized Study (LEVEL-AT)
Brief Title: LEft VEntricuLar Activation Time Shortening With Physiological Pacing vs Biventricular Resynchronization Therapy
Acronym: LEVEL-AT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josep Lluis Mont Girbau (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Centro de Investigación Biomédica en Red Enfermedades Cardiovasculares (CIBERCV) (Unknown)
Responsible Party: Sponsor-Investigator, Josep Lluis Mont Girbau, Head of Arrhythmia Section. Professor of Cardiology, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEVEL-AT
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Physiological Pacing; Resynchronization Therapy
Keywords: Physiological pacing; Resynchronization therapy; Electrocardiographic imaging

STUDY DESIGN:
Intervention Model Description: Randomized, unicentric, simple blind.
Who Masked: Participant
Masking Description: The patient will be explained to be randomized to either of the two branches. The type of therapy applied will not be communicated to the patient. The follow-up will be the same in the two branches. During the visits it will not be said which therapy has been applied.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Physiological pacing (Experimental): Pacing the his-purkinje system.
  Crossover to biventricular CRT will be allowed in the following situations: failed physiological pacing lead implantation; high thresholds (>3.5V / 1ms); no shortening of QRS (shortening <20%) or failure to meet non-selective HBP criteria [Europace. 2019 Oct 9. doi: 10.1093/europace/euz275].
  Interventions: Device: Lead placed in the His-Purkinje system in order to achieve QRS shortening.
- Biventricular resynchronization therapy (Active Comparator): Pacing from the right ventricular and coronary sinus leads. Electrocardiographic optimization with fusion-optimized intervals.
  Crossover from biventricular CRT to physiological pacing will be allowed in the following situations: coronary sinus cannot be cannulated; no lateral or posterolateral branches; or phrenic stimulation.
  Interventions: Device: Lead is placed in a tributary of the coronary sinus.

INTERVENTIONS:
Device: Lead placed in the His-Purkinje system in order to achieve QRS shortening. — Physiologic pacing to achieve QRS shortening. If the patient has indication of stimulation (AV block), a backup lead will be implanted in the right ventricle. All patients will have a lead placed in the right atrium (except those that have permanent atrial fibrillation).
  Arms: Physiological pacing
Device: Lead is placed in a tributary of the coronary sinus. — Biventricular Resynchronization Therapy is the use of a pacemaker with two endocardial leads placed in the right atrium and right ventricle. The third lead is placed in a tributary of the coronary sinus.
  Arms: Biventricular resynchronization therapy

SUMMARY:
The LEVEL-AT Trial (LEft VEntricuLar Activation Time Shortening with Physiological Pacing vs Biventricular Resynchronization therapy: a randomized study) is a non-inferiority study that aims to determine if physiological pacing could decrease the left ventricular activation time compared with biventricular therapy.

DETAILED DESCRIPTION:
To date studies have showed that physiological pacing could get similar clinical and echocardiographic response to that obtained with biventricular therapy. Activation time shortening with permanent physiological pacing has not been studied.

This study will randomize 70 patients to a strategy of: biventricular pacing versus physiological pacing.

LEVEL-AT study will analyze the following parameters in the 2 groups: shortening of the QRS, activation time with electrocardiographic imaging, echocardiographic asynchrony and ventricular function and clinical parameters (NYHA functional class, mortality and heart failure hospitalization).

Clinical, electrocardiographic, echocardiographic and electrocardiographic imaging follow-up will be performed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* The patient must indicate their acceptance to participate in the study by signing an informed consent document.
* The patient must be ≥ 18 years of age.
* Left bundle branch block, QRS ≥130 and FEVI <=35% (Indication of cardiac resynchronization IA or IB ESC Guidelines). No indication of stimulation for AV block.
* Patients with indication of resynchronization therapy for ventricular dysfunction and indication of cardiac stimulation for AV block according to ESC Guidelines (IA ESC Guidelines).
* Non-left bundle branch block, QRS ≥150 and FEVI <=35% (Indication of cardiac resynchronization IIaB ESC Guidelines).

Exclusion Criteria:

* Myocardial infarction, unstable angina or cardiac revascularization during the previous 3 months.
* Pregnancy.
* Participating currently in a clinical investigation that includes an active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Left ventricular activation time. | 45 days
  Left ventricular activation time measured by eletrocardiographic imaging.

SECONDARY OUTCOMES:
QRS duration. | Implant, 6 months and 12 months.
  QRS duration (milliseconds) measured with a 12-lead ECG.
Left ventricular activation time. | 6 months and 12 months.
  Left ventricular activation time measured by eletrocardiographic imaging
Change in left ventricular function. | 6 months and 12 months.
  Left ventricular ejection fraction measured with Simpson method with echocardiography.
Change in end-systolic volume. | 6 months and 12 months.
  End-systolic volume measured with echocardiography.
Change in NYHA functional class. | 6 months and 12 months.
  NYHA functional class I, II, III, IV.
Hospitalization due to heart failure or mortality (combined endpoint). | 1 year.
  Hospitalization: patient hospitalization (yes/no) Mortality: mortality (yes/no)
Correction of septal flash | 15 days
  Correction of septal flash determined with echocardiography (M mode)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Tolosana, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Margarida Pujol Lopez, MD, Principal Investigator — Hospital Clinic of Barcelona; Lluis Mont Girbau, MD, PhD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Select, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pujol-Lopez M, Ferro E, Borras R, Garre P, Guasch E, Jimenez-Arjona R, Garcia-Ribas C, Doltra A, Niebla M, Carro E, Roca-Luque I, Guichard JB, Puente JL, Uribe L, Vazquez-Calvo S, Castel MA, Arbelo E, Porta-Sanchez A, Sitges M, Tolosana JM, Mont L. Stepwise application of ECG and electrogram-based criteria to ensure electrical resynchronization with left bundle branch pacing. Europace. 2023 Jun 2;25(6):euad128. doi: 10.1093/europace/euad128. PMID 37294671
- [Derived] Pujol-Lopez M, Jimenez-Arjona R, Garre P, Guasch E, Borras R, Doltra A, Ferro E, Garcia-Ribas C, Niebla M, Carro E, Puente JL, Vazquez-Calvo S, Invers-Rubio E, Roca-Luque I, Castel MA, Arbelo E, Sitges M, Brugada J, Tolosana JM, Mont L. Conduction System Pacing vs Biventricular Pacing in Heart Failure and Wide QRS Patients: LEVEL-AT Trial. JACC Clin Electrophysiol. 2022 Nov;8(11):1431-1445. doi: 10.1016/j.jacep.2022.08.001. Epub 2022 Oct 26. PMID 36424012